CLINICAL TRIAL: NCT03795155
Title: Prospective Genomics Initiative on Multiple Synchronous Lung Cancer (PGI-MSLC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RenJiH-2018-056
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Multiple Synchronous Lung Cancers (MSLCs)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study is to characterize the genomic landscape and genetic heterogeneity of multiple synchronous lung cancer (MSLC) in correlation with comprehensive clinical, histopathological and medical imaging information, in order to improve disease diagnosis and tailored treatment for MSLC patients.

DETAILED DESCRIPTION:
* To initiate a prospective registry of MSLC patients with high-quality clinical samples and detailed medical data.
* To define the clonal relationship, genomic landscape and potential driver alterations of MSLC using whole-genome sequencing.
* To determine the intrapatient and intratumor genetic heterogeneity of MSLC.
* To correlate molecular features with clinical parameters and patient outcome.
* To serve as a continuous infrastructure for a large variety of research purposes including: A. Diagnostic research B. Prognostic research C. Biological research D. Interventional trial design testing new therapies in MSLC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Confirmed diagnosis of multiple synchronous lung cancers (MSLCs) without metastatic disease
* Signed informed consent

Exclusion Criteria:

* Medical or psychiatric condition that would preclude informed consent
* History of known high-risk infections
* With metastatic tumors except lung

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of multiple synchronous lung cancers (MSLCs)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Genomic characters of synchronous lessions in each MSLC patient | November 30, 2021
  Whole-genome sequencing reveals the mutation, copy number variation and structure variation of MSLCs. We will analysis the genomic characters of synchronous lesions in each MSLC patient.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Zhao, M.D., Principal Investigator — Ren Ji Hospital; Yujie Fu, Ph.D., Principal Investigator — Ren Ji Hospital; Guanglei Zhuang, Ph.D., Principal Investigator — Ren Ji Hospital
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma P, Fu Y, Cai MC, Yan Y, Jing Y, Zhang S, Chen M, Wu J, Shen Y, Zhu L, Chen HZ, Gao WQ, Wang M, Gu Z, Bivona TG, Zhao X, Zhuang G. Simultaneous evolutionary expansion and constraint of genomic heterogeneity in multifocal lung cancer. Nat Commun. 2017 Oct 10;8(1):823. doi: 10.1038/s41467-017-00963-0. PMID 29018192